CLINICAL TRIAL: NCT05956548
Title: Contrasting Lead Migration During Spinal Stimulation Trial Period Against Therapeutic Response - Evaluating Securement Methods During the Trial Period
Brief Title: Lead Migration During the Spinal Cord Stimulation Trial Period and Therapeutic Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Stephanie Jones, Principal Investigator, Augusta University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1994689
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Stimulator Trial Period, Neuromodulation Trial Period, SCS Trial Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: external securement of scs leads during the scs trial period — two groups- one group will have an anchor device used alone to secure the leads, the second group will have an anchor device with a suture to secure the leads

SUMMARY:
The goal of this clinical trial is to compare lead migration distance and therapeutic response for participants receiving a spinal cord stimulator during the trial period. Of note- scs trial period is a procedure name, not to be confused with this clinical trial study.

The main question[s] it aims to answer are:

* Is there a difference in migration distance and/or rate for those with external leads secured by an anchor device versus and anchor device with suture?
* How does participant activity levels during the trial period compare to migration rates? ° Does the temperature, heat index, and humidity during the trial period impact migration rates? Participants will come in for the scs trial procedure as normal. They will be asked to complete an activity survey upon return to the clinic for lead pull after the scs trial. They will also have an additional image upon return to the clinic to document lead position prior to lead pull.

Researchers will compare two groups- those with securement via anchor and those with securement via anchor and suture to see if there is an impact on therapeutic effect (percentage of pain relief) form the scs trial.

ELIGIBILITY:
Inclusion Criteria:

Adults ages 18 and over without a failed spinal stimulation trial or implant will be accepted into the study. Patients must have a diagnosis of chronic back pain and must be patients of the identified anesthesiologists and have their procedures performed at AUHS pain clinic.

Exclusion Criteria:

Patients will be excluded if they have a history of local anesthetic allergy (lidocaine), current skin infections at the procedure site, or a diagnosis of diaphoresis/ secondary hyperhidrosis (chronic over sweating).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-05-14 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Response | SCS trial periods are 3-6 days at our facilty.
  % of pain relief achieved by the participant during the SCS trial period
Lead position changes (migration) | the last day of the trial period which could be day 3 up to day 6, depending on length
  final location of the SCS leads at the end of the scs trial period, as seen on imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jeane Silva, PhD, Study Chair — Augusta University; Stephanie C Jones, Grad Student, Principal Investigator — Augusta University
Locations (1):
- Augusta University Health System Pain Clinic, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided